CLINICAL TRIAL: NCT05554536
Title: Evaluation of Regional Lung Mechanics in Obese Patients Undergoing Laparoscopic Surgery Using Electrical Impedance Tomography
Brief Title: Evaluation of Regional Lung Mechanics in Obese Patients Undergoing Laparoscopic Surgery
Acronym: OBESE-EIT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi di Ferrara (Other)
Responsible Party: Principal Investigator, Savino Spadaro, Clinical Professor, Università degli Studi di Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OBESE-EIT
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Obesity; Mechanical Ventilation Pressure High; Intraoperative Respiratory Injury
Keywords: EIT; Obesity; Laparoscopy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm intervention (Other): All patients will undergo a PEEP titration trial in each surgery step (before pneumoperitoneum, during pneumoperitoneum, after pneumoperitoneum). The PEEP titration trial will be done in steps of 2 cmH2O, starting from clinical PEEP 16 cmH2O and ending to PEEP 6 cmH2O. Each PEEP level will be kept for 2 minutes. The PEEP titration trial will be stopped in case of haemodynamic instability or severe desaturation (Spo2 < 92%). Each PEEP titration trial will be recorded using Electrical impedance tomography (EIT).
  Interventions: Procedure: PEEP titration trial

INTERVENTIONS:
Procedure: PEEP titration trial — PEEP trial, starting from clinical PEEP 16 cmH2O and ending at PEEP 6 cmH2O. The PEEP trial will be stopped for haemodynamic instability (defined as arterial pressure < 80 mmHg and /or heart rate > 150 bpm) or desaturation (defined as SpO2 < 92%).

SUMMARY:
This study will evaluate what is the impact of laparoscopy and Trendelenburg position on lung regional ventilation distribution in obese patients, focusing on the differences between the different phases of surgery.

DETAILED DESCRIPTION:
Electrical impedance tomography (EIT) is a non invasive monitoring technique that allows to evaluate the regional distribution of ventilation. EIT has been used in different contexts, such as acute respiratory failure or intraoperative ventilation settings. Obesity, by increasing intrabdominal pressure, may reduce functional residual capacity after anesthesia and therefore require a more aggressive intraoperative ventilatory setting. In addition, laparoscopy, by increasing the volume of the abdomen, further pushes the diaphragm and increase the probability of lung collapse.

The aim of the current study is to describe the effect of 1) anesthesia and of 2) laparoscopy and trendelenburg position on regional ventilation distribution. Moreover, the investigators will evaluate if the best ventilatory parameters set after anesthesia induction are confirmed also when the condition changes (i.e. during pneumoperitoneum and trendellenburg).

Finally, the investigators will explore if the different parameters which can be provided by EIT agree in suggesting the best level of positive-end expiratory pressure in both moments of surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18-90 years
* Body mass index > 30 kg/m2
* Major surgery
* Predicted duration of surgery > 2 hours
* Predicted presence of invasive arterial pressure monitoring

Exclusion Criteria:

* emergency surgery
* Refuse to participate from patient
* presence of Implantable cardiac device or pacemaker
* thoracic wounds
* thoracic surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Best Positive end-expiratory pressure - Laparoscopy variability | Difference between the best PEEP after anesthesia induction and during pneumoperitoneum
  The primary outcome will be the best PEEP found using the PEEP titration trial.

SECONDARY OUTCOMES:
Best Positive end-expiratory pressure - EIT variability | After anesthesia induction, during pneumoperitoneum, end of surgery
  Secondary outcome will be to compare the different values of best PEEP provided by several parameters of EIT to evaluate if the overlap.

CONTACTS AND LOCATIONS:
Overall Officials: Savino Spadaro, MD, PhD, Study Director — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero Universitaria Sant'Anna, Ferrara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erlandsson K, Odenstedt H, Lundin S, Stenqvist O. Positive end-expiratory pressure optimization using electric impedance tomography in morbidly obese patients during laparoscopic gastric bypass surgery. Acta Anaesthesiol Scand. 2006 Aug;50(7):833-9. doi: 10.1111/j.1399-6576.2006.01079.x. PMID 16879466
- [Background] Zhu C, Yao JW, An LX, Bai YF, Li WJ. Effects of intraoperative individualized PEEP on postoperative atelectasis in obese patients: study protocol for a prospective randomized controlled trial. Trials. 2020 Jul 6;21(1):618. doi: 10.1186/s13063-020-04565-y. PMID 32631414
- [Background] Spinelli E, Mauri T, Fogagnolo A, Scaramuzzo G, Rundo A, Grieco DL, Grasselli G, Volta CA, Spadaro S. Electrical impedance tomography in perioperative medicine: careful respiratory monitoring for tailored interventions. BMC Anesthesiol. 2019 Aug 7;19(1):140. doi: 10.1186/s12871-019-0814-7. PMID 31390977
- [Background] de Castro Martins T, Sato AK, de Moura FS, de Camargo EDLB, Silva OL, Santos TBR, Zhao Z, Moeller K, Amato MBP, Mueller JL, Lima RG, de Sales Guerra Tsuzuki M. A Review of Electrical Impedance Tomography in Lung Applications: Theory and Algorithms for Absolute Images. Annu Rev Control. 2019;48:442-471. doi: 10.1016/j.arcontrol.2019.05.002. Epub 2019 May 17. PMID 31983885
- [Derived] Scaramuzzo G, Priani P, Ferrara P, Verri M, Montanaro F, La Rosa R, Cammarota G, Volta CA, Spadaro S. Longitudinal changes of electrical impedance tomography-based best PEEP in obese patients undergoing laparoscopic surgery: A prospective physiological study. Anaesth Crit Care Pain Med. 2025 Sep;44(5):101569. doi: 10.1016/j.accpm.2025.101569. Epub 2025 Jun 13. PMID 40518045